CLINICAL TRIAL: NCT02818543
Title: An Open-Label, Single Ascending Dose Study To Evaluate The Pharmacokinetic Profile, Safety and Tolerability of Orally Administered LYC-30937 in Subjects With Active Ulcerative Colitis
Brief Title: Safety and Pharmacokinetic Study of LYC-30937 in Subjects With Active Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lycera Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: LYC-30937-1002
Record Dates: First submitted 2016-03-30; First posted 2016-06-29 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): LYC-30937 25 mg single oral dose
  Interventions: Drug: LYC-30937
- Cohort 2 (Experimental): LYC-30937 100 mg single oral dose
  Interventions: Drug: LYC-30937

INTERVENTIONS:
Drug: LYC-30937

SUMMARY:
The purpose of this study to assess the pharmacokinetic profile in patients with active ulcerative colitis and compare it to the experience in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Active ulcerative colitis defined as a Mayo endoscopy score of ≥ 2 despite therapy.
* Male or female age 18 to 75
* May be receiving a therapeutic dose of an oral 5-amino salicylic acid compound or oral corticosteroid therapy

Exclusion Criteria:

* Current anti-tumor necrosis factor use
* Current immunosuppressant use (Note: this does not include corticosteroid use)
* Subjects with only distal active disease (i.e. proctitis)
* Clinically significant active infection
* Known bleeding disorder, a risk of bleeding or hypercoagulable disorders in which an anticoagulant is required
* History of malignancy within the last 5 years except non-melanoma skin cancer or cervical carcinoma in situ
* Clinically significant lab abnormalities (i.e. liver function abnormalities, renal insufficiency, abnormal absolute neutrophil count or hemoglobin)
* History of colon resection
* Any other investigational therapy or investigational biologics use within 8 weeks of investigational medicinal product administration

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | up to 48 hours
  Measure specified pharmacokinetic parameters pre-dose and out to 48 hours post-dose
Time to maximum observed plasma concentration (Tmax) | up to 48 hours
  Measure specified pharmacokinetic parameters pre-dose and out to 48 hours
Percentage of estimated Area Under the Curve (0-inf) | up to 48 hours
  Measure specified pharmacokinetic parameters pre-dose and out to 48 hours

SECONDARY OUTCOMES:
Treatment emergent adverse events (TEAEs) | 7 days post-dose
  TEAEs will be listed and summarized by dose and overall
Clinical laboratory data | 7 days post-dose
  Clinical laboratory data will be listed with flagging of values outside the normal range
Vital signs | 7 days post-dose
  descriptive statistics will be provided to summarize vital signs and changes from baseline by dose at each scheduled time
12-Lead Electrocardiogram (ECG) | 7 days post-dose
  Descriptive statistics will be provided to summarize ECG parameters

CONTACTS AND LOCATIONS:
Locations (2):
- Hungary (2):
  - DRC Ltd., Balatonfüred
  - PRA Magyarorszag Kft, Budapest

IPD SHARING:
Plan to Share IPD: No